CLINICAL TRIAL: NCT02832739
Title: Exploring Acceptance and Outcomes of an ICT-based Self-management Support System for Community-dwelling Older Adults With Chronic Diseases and Informal Caregivers: USECARE Study Protocol
Brief Title: Exploring Acceptance and Outcomes of an Online-based Self-management Support System in Chronic Illness
Acronym: USECARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assuta Medical Center (Other)
Collaborators: Norwegian Centre for Integrated Care and Telemedicine (NST) (Unknown); Open-Evidence c/o Universitat Oberta de Catalunya (Unknown); Institute for Health and Consumer Protection c/o University of Oslo, Faculty of Medicine (Unknown); European Medical Network EMN AG (Unknown)
Responsible Party: Principal Investigator, Jacob Gindin, Director Geriatric Services, Assuta Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IFI.2014.0056
Record Dates: First submitted 2016-06-08; First posted 2016-07-14 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Chronic Heart Failure; Diabetes Mellitus; Chronic Obstructive Pulmonary Disease; Special Orthopaedic Co-Morbidity After Hip/Knee Replacement
Keywords: Technology acceptance; Usability; eHealth; self-management support in chronic illness; prevention; Special Orthopaedic Co-Morbidity after hip/knee replacement
MeSH Terms: conditions — Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENACA - self-management support system (Experimental): Use of enhanced SENACA - ICT based self-management support system prototype by study participants at home for 75-100 days
  Interventions: Device: SENACA - ICT based self-management support system

INTERVENTIONS:
Device: SENACA - ICT based self-management support system — SENACA - ICT based self-management support system is a structured self-management support system with several interacting components, combining tele-monitoring devices and a solution for personalised health plans. ==> www.senaca.ch

SUMMARY:
The aim of the USECARE project is to improve and test SENACA, an ICT-based self-management support system for chronically ill patients and informal caregivers. 60 end-users will be instructed to use SENACA for approx. 3 months (in Israel and Norway). Amongst others, clinical and behavioural outcomes will be recorded. Additionally, SENACA's usability will be evaluated to determine its potential future scalability.

DETAILED DESCRIPTION:
In Switzerland, SENior health ACAdemy (SENACA, www.senaca.ch) has been developed by the European Medical Network EMN.

SENACA is a structured self-management support system with several interacting components, combining tele-monitoring devices and a solution for personalised health plans. This online support system's usability, the behaviour change techniques it builds on, modes of delivery and its effects on health-related behaviour, clinical and Quality-of-Life outcomes will be established in a larger group of end-users.

Testing the usability of SENACA and practical effectiveness of this intervention is the goal of this multi-national project USECARE (www.usecare.eu).

SENACA will be implemented in two countries (Israel and Norway ) via field test with community-dwelling older adults living with chronic conditions (i.e. diabetes, COPD, chronic heart failure) and their informal caregivers.

Key element of USECARE is a field-test including a study based upon pre-experimental design with three time point measurements and a pre-usability round. Multiple methods will be used to evaluate the usability and to observe clinical and process parameters before, during and after the implementation of the enhanced SENACA prototype.

All of the results combined will provide an insight into the end-user experience, usage pattern, usability perception and potential added value of the enhanced SENACA prototype for chronic disease management in the participating countries.

ELIGIBILITY:
Inclusion community-dwelling older adults (primary end-users):

* receive medical care for one or more of the following chronic diseases in hospital settings and outpatient clinics:

  1. Chronic Heart Failure (CHF, New York Heart Association NYHA IIIIIa);
  2. Diabetes Mellitus (DM, 6< HbA1c<9),
  3. Chronic Obstructive Pulmonary Disease (COPD, GOLD I-II)
  4. Special Orthopaedic Co-Morbidity (SOCM, after elective hip or knee replacement, health status temporarily destabilized respectively challenged, increased monitoring and formal/informal care).
* having support of an informal caregiver that is aged 18 years or older
* aged 50 years and older (primary end-users)

Exclusion community-dwelling older adults (primary end-users):

* known illiteracy (reading and writing difficulties)
* lack of local language proficiency
* current major mental illness of moderate to severe level
* major acute illness or surgery in past 3 months (except elective hip / knee surgery for patients with SOCM)
* participation in another intervention study

Inclusion informal caregivers (secondary end-users):

* aged 18 years or older
* named by primary end-user as designated informal caregiver providing physical, emotional and/or social support for him or her

Both inclusion criteria primary and secondary end-users:

* written informed consent
* adequate functional, sensory and cognitive abilities to use the SENACA system

Both exclusion criteria primary and secondary end-users:

* does not have a stable address of residence
* no internet/computer access
* inability to handle ICT-devices due to cognitive or functional disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-08-31 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Level of and potential changes in technology acceptance in participants | Up to three months
  Technology acceptance (usability) of system is measured by assessing participants' intention to use, perceived ease of use, perceived usefulness, technology experience, preference in using technology, errors, and user satisfaction. Instruments used are: Technology Acceptance Model (TAM), Post-Study System Usability Questionnaire (PSSUQ), all self-reported questionnaires. In addition, system errors will be reported (number and type of problems).

SECONDARY OUTCOMES:
Level of and potential changes in selected clinical outcomes of participants : BMI, weight, fasting glucose as well as HbA1c levels (sample) | Up to three months
  Changes in selected clinical outcomes will be assessed with automated measurements via the intervention devices concerning body fat (fat proportion of body in %), body weight (in kg), blood pressure (systolic/diastolic in mmHg), pulse (per minute), SpO2 (in %) and fasting glucose (mmol). In Norway sample laboratory test will be conducted to determine levels of cholesterols (HDL, LDL in mmol), triglyceride (in mmol), HbA1c (mmol) and BNP (pg/ml).
Level of and potential changes in health-related quality of life of participants assessed by EQ5D5L | Up to three months
  Use of EQ-5DL a standardised instrument to measure health outcome and health-related quality of life.
Level of and potential changes in uptake and usage of the SENACA intervention by participants | Up to three months
  Automated recording of relative frequency of usage of SENACA's modules (usage of single components that are not mandatory), adherence to SENACA (Number of days within program from initiation to discontinuation (time to event), errors of system during intervention (number and type of technical problems occurring)
Level of and potential changes in self-efficacy of participants | Up to three months
  Measured with the Stanford Self-efficacy for managing chronic disease scale (SES6)
Level of and potential changes in health-related behaviour: nutrition & alcohol consumption, smoking, physical activity | Up to three months
  Self-reported questionnaires on weekly unit consumption (nutrition/alcohol), exercise (in Norway) and walking (minutes or hours/week), smoking behaviour (tobacco products, consumption per day), alcohol (units/week).Physical activity will be recorded automatically via pedometer (device).
Level of and potential changes in eHealth Literacy in participants | Up to three months
  eHealth Literacy is defined as the ability to read, use computers, search for information, understand health information, and put it into context.The eHealth Literacy Scale (eHEALS) as an 8-item measure will be used (self-reported questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Frank Larsen, MA, Study Chair — Norwegian Centre for Integrated Care and Telemedicine
Locations (2):
- Assuta Medical Center, Tel Aviv, Israel
- University Hospital North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No